CLINICAL TRIAL: NCT05798741
Title: Hardware Removal After ORIF of Ankle Fractures: A Randomized Trial
Brief Title: Hardware Removal After ORIF of Ankle Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00026
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Hardware Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hardware removal (Experimental): hardware removal
  Interventions: Procedure: Hardware removal
- hardware retaining (No Intervention): Patients that retain their hardware

INTERVENTIONS:
Procedure: Hardware removal — The surgery of hardware removal after an ORIF of an ankle fracture
  Arms: Hardware removal

SUMMARY:
Ankle fractures account for 10 % of fractures in the adult population. A part of patients (40%) is treated surgically. After healing of the fractures, about one year after the operation, a surgery is often performed to remove the hardware in order to diminish pain. If this surgery is necessary is debated in the literature.

The aim of our study is to evaluate the outcome of hardware removal surgery after a surgery of the ankle for a fracture. For that, we will perform do a controlled randomized trial with two arms: one arm includes the participants who will have a hardware removal and the other arm will not have a surgery.

Outcome parameters are the patients reported outcome and pain related disability. They will be assessed by the questionnaires FAAM score (Foot and Ankle Ability Measure) and PDI (Pain Disability Index) at the beginning and at the end of the study, at six months. The third outcome parameter will be the complication rate after an anklehardware removal surgery, which will be assessed through the Ernst-Ssink classification.

DETAILED DESCRIPTION:
The study consists of a prospective multicentric parallel two-arm randomised non-blinded study, conducted at the HFR and RHNe (level of evidence II).

The planned intervention is the following: after an ORIF of the ankle, patients have a follow-up. At the 12- month control, we ask eligible patients if they want to participate to the study. If they agree, they are randomised to treatment recommendations in one of two groups: conservative or surgical. The patients may follow or not the recommendations; not following the recommendations does not exclude them from the study. Patients of both groups will fill out FAAM and PDI questionnaires at 12 and 18 months after the 1st operation. Patients in the surgical group will have a hardware removal surgery. It is a very common operation consisting of hardware removal that is done ambulatory by the orthopaedic surgeons specialized in foot and ankle surgery. Operated patients will have the usual postoperative follow-up (6 weeks, 3 months and 6 months postoperative) and all complications will be recorded and classified according to the Ernst-sink classification

ELIGIBILITY:
Inclusion Criteria:

* >18 y.o
* Operative treatment of ankle/foot fractures at HFR or RHNe:
* Ankle fractures: bi-malleolar and tri-malleolar fractures or equivalent
* FAAM score >5%, <95%
* Patient expected to complete length of study
* Patient with sufficient cognitive and linguistic ability in order to participate in the study.
* Operable patients (ASA score ≤3)

Exclusion Criteria:

* Absolute indications for HR: infection/malunion/allergy to metal/refracture
* Ankle fractures that are not listed in the criteria above
* Patient treated for a fracture at the same foot/ ankle before
* Patient with fracture of two different regions of the foot/ankle
* Patient treated for the fracture outside of HFR and RHNe
* Patient non ambulating before time of injury
* Patients having diabete,
* immunocompromised under chemotherapy,
* Peripheral artery disease stade IV
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
patient reported outcome after an ankle hardware removal | 6 months
  FAAM score (Foot and Ankle Ability Measure). FAAM subdivided in AVQ scale(84 points) and Sport scale (32 points). The higher is a better outcome.

SECONDARY OUTCOMES:
pain-related disability after an ankle hardware removal | 6 months
  PDI (Pain Disability Index). Total of 70 points. The higher means a worse outcome.
complication rate after an ankle hardware removal surgery | 6 months
  Ernst-sink classification